CLINICAL TRIAL: NCT05786144
Title: Vestibular Schwannoma Stem Cell Organoids
Brief Title: Vestibular Schwannoma Organoids
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Schwannoma organoids
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In standard of care regularly planned surgery, tissue will be obtained from patients who are suspicious for having vestibular Schwannoma (on MRI). The tissue that remains after the pathologist gathered sufficient for analysis, the remaining tissue is used for creating tumour stem cell organoids.

DETAILED DESCRIPTION:
This project constitutes scientific research since the presence of tumor stem cells has not been shown in schwannoma before. Secondly the organoid model has not yet been described for VSs. The correlation between effect in schwannoma organoids and in patients has to be evaluated but can proof to be very valuable since it has been shown in a number of tumors. The tumor tissue will be acquired during regularly planned surgery. The tissue that is used is what is left after sufficient material has been sent to the pathologist to make the diagnosis. So the tissue that is used is removed routinely during surgery, but instead of banking it at the pathology department, it is used for the research project. Blood samples that can be used to compare normal DNA to tumor cells DNA will be acquired from central lines that are routinely placed during these procedures, so no additional interventions will be done in acquiring the tissue and blood for this study.

ELIGIBILITY:
Inclusion Criteria:

* MRI with suspicion for vestibular schwannoma
* Indication for surgery in the skull base committee
* 18 years or older

Exclusion Criteria:

* Refusal to participate
* Younger than 18 years
* Incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a supsicion for vestibular schwannoma on an MRI for which surgery was indicated (approximately 10 per year in Maastricht).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | 10 years
  Feasibility to create organoids from schwannoma tumour tissue and make a "living" biobank of these tissues in the laboratory to study the resistance mechanisms towards treatments.

SECONDARY OUTCOMES:
Phenotype | 10 years
  Comparing the phenotypical profile of the vestibular schwannoma organoid to the phenotypical profile of the original tumour.
Genetic | 10 years
  Comparing the genetic profile of the vestibular schwannoma organoid to the genetic profile of the original tumour.
Epigenetic | 10 years
  Comparing the epigenetic profile of the vestibular schwannoma organoid to the epigenetic profile of the original tumour.
Proteomic | 10 years
  Comparing the proteomic profile of the vestibular schwannoma organoid to the proteomic profile of the original tumour.
Transcriptomic | 10 years
  Comparing the transcriptomic profile of the vestibular schwannoma organoid to the transcriptomic profile of the original tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Koos Hovinga, Principal Investigator — Maastricht University Medical Center; Marc Vooijs, MD, PhD, Principal Investigator — Maastro
Locations (2):
- Netherlands (2):
  - Maastro, Maastricht, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg